CLINICAL TRIAL: NCT01511692
Title: A 4 Week Single Center, Double-dummy, Randomised Double-blind, Balanced Incomplete Latin Square Design Study to Evaluate the Effects of Liraglutide on Appetite in Subjects With Type 2 Diabetes Compared to Glimepiride and Placebo
Brief Title: Effect of Liraglutide Compared to Glimepiride on Appetite in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1589; 2006-000377-30 (EudraCT Number)
Record Dates: First submitted 2012-01-12; First posted 2012-01-19 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lira --> placebo (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- Placebo --> glim (Placebo Comparator)
  Interventions: Drug: placebo; Drug: glimepiride
- Glim --> lira (Active Comparator)
  Interventions: Drug: liraglutide; Drug: glimepiride

INTERVENTIONS:
Drug: liraglutide — 1.8 mg/day injected subcutaneously for 4 weeks
  Arms: Glim --> lira; Lira --> placebo
Drug: placebo — Liraglutide placebo, injected subcutaneously for 4 weeks
  Arms: Lira --> placebo
Drug: placebo — Glimepiride placebo, dose individually adjusted, administered orally for 4 weeks
  Arms: Placebo --> glim
Drug: glimepiride — Dose individually adjusted, administered orally for 4 weeks
  Arms: Glim --> lira; Placebo --> glim

SUMMARY:
This trial is conducted in Europe and Oceania. The aim of this trial is to assess the effects of liraglutide on energy intake in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Diet-treated subjects and/or subjects with type 2 diabetes in OAD (oral anti-diabetic drug) mono-therapy
* HbA1c for diet-treated subjects: HbA1c between 6.5-10.0% (both inclusive) and for OAD treated subjects: HbA1c between 6.5-9.5% (both inclusive)
* Body mass index (BMI) between 27-40 kg/m^2 (both inclusive)
* Subjects should have a stable body weight for at least 3 months prior to screening (as documented by a weight within 3 to 6 months, prior to screening that is within 15% of the screening weight)
* Euthyroid subjects
* Subjects should be unrestrained eaters

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Impaired liver function
* Impaired renal function
* Cardiac problems
* Uncontrolled treated/untreated hypertension
* Known or suspected allergy to trial products or related products
* Use of any drug (except for OADs), which in the investigator's opinion could interfere with the subject's glucose level or body weight
* Active hepatitis B and/or active hepatitis C
* Positive HIV (human immunodeficiency virus) antibodies
* Known or suspected abuse of alcohol or narcotics
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, cola drinks, chocolate) as judged by the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The energy intake at a standardised buffet meal with a preload paradigm quantified using Foodworks 2.10

SECONDARY OUTCOMES:
The energy intake at a standardised buffet meal without a preload paradigm quantified using Foodworks 2.10
Macronutrient distribution of food consumed at a standardised buffet meal with a preload paradigm quantified using Foodworks 2.10
Macronutrient distribution of food consumed at a standardised buffet meal without a preload paradigm quantified using Foodworks 2.10
Total duration of eating at the buffet meal (satiation)
Weight
Waist circumference
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Adelaide, South Australia, Australia
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Horowitz M, Flint A, Jones KL, Hindsberger C, Rasmussen MF, Kapitza C, Doran S, Jax T, Zdravkovic M, Chapman IM. Effect of the once-daily human GLP-1 analogue liraglutide on appetite, energy intake, energy expenditure and gastric emptying in type 2 diabetes. Diabetes Res Clin Pract. 2012 Aug;97(2):258-66. doi: 10.1016/j.diabres.2012.02.016. Epub 2012 Mar 24. PMID 22446097
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com